CLINICAL TRIAL: NCT04944667
Title: Use of Virtual Reality for Procedural Planning of Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: Use of Virtual Reality for Procedural Planning of Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Collaborators: Techer Team SL. Valencia. Spain (Unknown)
Responsible Party: Principal Investigator, Eduard Permanyer, Md,PhD, Centro Medico Teknon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cardiac Surgery CentroMT
Record Dates: First submitted 2021-06-09; First posted 2021-06-29 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVR standard (Other): TAVR planning evaluated without VR and TAVR planning after VR analysis
  Interventions: Diagnostic Test: TAVR planning

INTERVENTIONS:
Diagnostic Test: TAVR planning — TAVR planning without VR vs after VR

SUMMARY:
This study sought to evaluate the impact of Virtual Reality (VR) tools in procedural planning of transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
A prospective study involving 11 patients referred for TAVR was conducted. A multidetector computed tomography (MDCT) was used to acquire and segment the anatomy of the access route and landing zone. From the information obtained with the MDCT in DICOM format, the investigators built a virtual platform (VisuaMed, Teacher Team. Valencia. Spain) that contains all the clinical information of the patients and a virtualized model of their anatomy. Wearing VR devices, the professional was able to "walk inside " the anatomy in an interactive and immersive way. Decisions after the evaluation of routine clinical images were compared with those after experience with VR models and intraprocedural findings.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis considered for TAVR procedure at a single Institution

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
TAVR procedure planning (prosthesis size, implant technique requirements, potential risks) | Baseline
  Does the TAVR procedure planning change after VR?

CONTACTS AND LOCATIONS:
Locations (1):
- CentroMT (Centro Médico Teknon), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No